CLINICAL TRIAL: NCT06691438
Title: Evaluation of the Effect on Pain of Attentional Diversion Associated with Hypnotic Induction by Virtual Reality (VRH) in Perioperative Prostate Biopsies Under Local Anesthesia: Prospective Randomized and Controlled Trial
Brief Title: Evaluation of the Effect on Pain of Attentional Diversion Associated with Hypnotic Induction by Virtual Reality (VRH) in Perioperative Prostate Biopsies Under Local Anesthesia:
Acronym: HYPNOSURG-VR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, EssaiClinique_HYPNOSURG-VR, Professeur, University Hospital, Grenoble
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EssaiClinique_HYPNOSURG-VR
Record Dates: First submitted 2024-10-21; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Prostate Biopsy
Keywords: Sedation; Pain; Hypnosis; Virtual Reality
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The maximum value of the pain will be collected by the research associate or the coordinating nurse who will be blinded to the randomization arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- prostate biopsies without virtual reality hypnosis headset (Active Comparator): Biopsies are performed according to current recommendations
  Interventions: Device: prostate biopsy
- prostate biopsies with virtual reality hypnosis headset (Experimental): Patient wearing a virtual reality headset put in place in the transfer room 15 minutes before the procedure and maintained throughout the procedure.
  Interventions: Device: prostate biopsy

INTERVENTIONS:
Device: prostate biopsy — prostate biopsies with virtual reality hypnosis headset
  Other Names: experimental

SUMMARY:
The primary objective of the study is to prospectively compare perioperative pain assessed in patients undergoing targeted prostate biopsies, either transrectally or transperineally, under local anesthesia with or without a virtual reality hypnosis headset. The study was sized based on a mean pain reduction of 1.5 points on a numerical scale (0-10 NAS), with an estimate of procedure-related pain of 4.0 on the NAS scale.

DETAILED DESCRIPTION:
Prospective comparison of pain during the procedure assessed in patients treated for prostate biopsies under local anesthesia with or without a virtual reality headset.No additional examination will be performed in addition to the conventional management of a biopsy except for the fitting of the headset for patients randomized to the "with virtual reality headset" group.

Patients will be randomized on the same day of the procedure into one of the two study groups.

A single follow-up visit will be performed postoperatively 1 month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are candidates for ultrasound-guided prostate biopsies under local anesthesia, via transperineal or transrectal route
* Patient having signed informed consent

Exclusion Criteria:

* Patient suffering from blindness or any other visual handicap that contraindicates the use of the headset
* Deaf or hard of hearing patients
* Patients suffering from epilepsy and/or mental deficiency, and/or disorders of higher functions
* Psychotic patients
* Claustrophobic patients or those who cannot tolerate a mask over their eyes
* Refusal of local anesthesia
* Protected person (art. L1121-5 to L1121-8 of the CSP)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 130 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
To prospectively compare perioperative pain assessed in patients undergoing targeted prostate biopsies, transrectally or transperineally, under local anesthesia with or without a virtual reality hypnosis headset. | after the procedure
  maximum pain felt during the procedure on a numerical EN scale, ranging from 0 (no pain) to 10 (extreme pain). The values will be collected directly at the end of the procedure.

SECONDARY OUTCOMES:
Pain after the procedure | when leaving the hospital
  Numerical scale 0-10 of pain upon discharge from the hospital
Stress during the procedure | after the procedure
  Numerical stress scale from 0 to 10 upon arrival of the patient, and 15 minutes after the procedure
Immersion during hypnosis | at the procedure
  Immersion scale from 0 to 10 during hypnosis
Evaluation of the nociceptive response to painful stimuli | during the procedure
  Heart rate variability (= HRV) on the ECG trace (in milliseconds)
Satisfaction with the procedure | after the procedure
  Desire to repeat this method of anesthesia in the event of an iterative procedure versus general anesthesia (yes/no)
Duration of the procedure | after the procedure
  Duration of the procedure in minutes (time between the start of the procedure and the end of the procedure by the surgeon)
Length of stay in hospital / outpatient care | at 1 month
  Length of stay in day hospital or outpatient care, in minutes (Time leaving the room - Time entering the room)
Success of biopsies | at 1 month
  Number of biopsies performed/planned (ratio), achievement of the MRI target (Yes/no)
Need for general anesthesia | after the procedure
  Rate of need for general anesthesia (in %)
Pain upon returning home the same evening and on D1 | after procedure, at 1 day after procedure
  Numerical pain scale 0-10 on returning home the same evening and on D1 collected in the patient notebook
Adverse effects related to the procedure during one month | at 1 month
  Patient notebook for collecting adverse effects for 1 month
Qualitative assessment of the patient's experience | after the procedure
  Semi-directed interview directly after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gaelle GF FIARD, professor, Principal Investigator — university grenoble hospital
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No